CLINICAL TRIAL: NCT04658316
Title: The Influence of Age and Gender on Tongue Pressure and Swallowing Tongue Pressure
Acronym: IOPI
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202010017RINB
Record Dates: First submitted 2020-11-30; First posted 2020-12-08 (Actual); Last update posted 2022-08-08 (Actual); Status verified 2020-11

CONDITIONS: Swallowing Disorder
Keywords: Swallowing function; Age; Gender
MeSH Terms: conditions — Deglutition Disorders; Coitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- 20-39Years-old Male: Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure.
  Interventions: Behavioral: Iowa Oral Performance Instrument
- 40-59Years-old Male: Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure.
  Interventions: Behavioral: Iowa Oral Performance Instrument
- 60-79Years-old Male: Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure.
  Interventions: Behavioral: Iowa Oral Performance Instrument
- 20-39Years-old Female: Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure.
  Interventions: Behavioral: Iowa Oral Performance Instrument
- 40-59Years-old Female: Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure.
  Interventions: Behavioral: Iowa Oral Performance Instrument
- 60-79Years-old Female: Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure.
  Interventions: Behavioral: Iowa Oral Performance Instrument

INTERVENTIONS:
Behavioral: Iowa Oral Performance Instrument — Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure

SUMMARY:
The main topic of the research is to investigate the tongue's strength when swallowing. There has been much foreign literature on tongue strength. Iowa Oral Performance Instrument also has norms for reference, but the data are all taken from non-Asian people such as Caucasians. In this case, the credibility of the norms are decreased in domestic, and we also lack norm data of tongue strength when swallowing. Through the research, we can establish normative data belonging to the domestics, provide usable data for domestic researchers and clinical staff, and explore whether there are differences in age and gender in data between Taiwanese and foreigners.

DETAILED DESCRIPTION:
Swallowing refers to the process by which food enters the stomach from the mouth. It is the physiological mechanism by which humans take in water and nutrients. It is a vital activity for individual survival. The physiological mechanism of swallowing has four major stages, oral preparation, oral cavity, pharynx, and esophagus. Each stage has its physiological mechanism, which depends on the different nerve and muscle structures. In the oral stage, our tongue plays an important role. Whether in the formation or transition of the food bolus, it must rely on the tongue to perform its normal functions. The main topic of the research is to explore the strength of the tongue when swallowing. The purpose is to discuss the influence of gender and age on swallowing tongue pressure. We expect to recruit 80 subjects and divide them into three groups according to their age: 20 to 39 years old, 40 to 59 years old, and 60 to 79 years old, with 13 to 14 males and females in each group, using Iowa Oral Performance Instrument measures the subject's maximum tongue pressure, average swallowing tongue pressure, and the ratio of the maximum tongue pressure used when swallowing, to explore whether age and gender affect tongue strength when swallowing.

ELIGIBILITY:
Inclusion Criteria:

* Aged twenty and above.

Exclusion Criteria:

* Based on self-representation, has the disease of the nervous system, included stroke, brain trauma, Parkinson's disease, dementia, etc.
* Based on self-representation, has head and neck cancers.
* Based on self-representation, had any history of swallowing disorders.
* Based on self-representation, has obvious cognition impairment or language disorder that will affect measure procedure.

Ages: 20 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Based on gender identity.
Study Population: Healthy adult.
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Iowa Oral Performance Instrument | immediately after the intervention/procedure/surgery
  Use Iowa Oral Performance Instrument to measure tongue pressure and swallowing tongue pressure of subject, in order to establish Taiwan's data.

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Chun Chih, Doctoral, Study Director — Chung Shan Medical University, Taiwan
Locations (1):
- National Taiwan University hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided
Undecided.

REFERENCES:
- [Background] 張家臻, 陳惠櫻, 李蕙蓉, 林宗豪, 謝佩君, 張雁雲, & 邱麗玲. (2018). 國 際吞嚥困難飲食標準中文繁體版本. 亞東學報, (38), 1-18.
- [Background] Adams V, Mathisen B, Baines S, Lazarus C, Callister R. A systematic review and meta-analysis of measurements of tongue and hand strength and endurance using the Iowa Oral Performance Instrument (IOPI). Dysphagia. 2013 Sep;28(3):350-69. doi: 10.1007/s00455-013-9451-3. Epub 2013 Mar 7. PMID 23468283
- [Background] Alsanei, W. A. S. (2015). Tongue Pressure-A Key Limiting Aspect in Bolus Swallowing (Doctoral dissertation, University of Leeds).
- [Background] Crow HC, Ship JA. Tongue strength and endurance in different aged individuals. J Gerontol A Biol Sci Med Sci. 1996 Sep;51(5):M247-50. doi: 10.1093/gerona/51a.5.m247. PMID 8808997
- [Background] Logemann, J. A. (1998). Evaluation and Treatment of Swallowing Disorders (2nd ed.). Austin, TX: Pro-Ed.
- [Background] Park JS, You SJ, Kim JY, Yeo SG, Lee JH. Differences in orofacial muscle strength according to age and sex in East Asian healthy adults. Am J Phys Med Rehabil. 2015 Sep;94(9):677-86. doi: 10.1097/PHM.0000000000000230. PMID 25415391
- [Background] Robinovitch SN, Hershler C, Romilly DP. A tongue force measurement system for the assessment of oral-phase swallowing disorders. Arch Phys Med Rehabil. 1991 Jan;72(1):38-42. PMID 1985622
- [Background] Robbins J, Kays SA, Gangnon RE, Hind JA, Hewitt AL, Gentry LR, Taylor AJ. The effects of lingual exercise in stroke patients with dysphagia. Arch Phys Med Rehabil. 2007 Feb;88(2):150-8. doi: 10.1016/j.apmr.2006.11.002. PMID 17270511
- [Background] Stierwalt JA, Youmans SR. Tongue measures in individuals with normal and impaired swallowing. Am J Speech Lang Pathol. 2007 May;16(2):148-56. doi: 10.1044/1058-0360(2007/019). PMID 17456893
- [Background] Vanderwegen J, Guns C, Van Nuffelen G, Elen R, De Bodt M. The influence of age, sex, bulb position, visual feedback, and the order of testing on maximum anterior and posterior tongue strength and endurance in healthy belgian adults. Dysphagia. 2013 Jun;28(2):159-66. doi: 10.1007/s00455-012-9425-x. Epub 2012 Sep 16. PMID 22983359
- [Background] Vitorino J. Effect of age on tongue strength and endurance scores of healthy Portuguese speakers. Int J Speech Lang Pathol. 2010 Jun;12(3):237-43. doi: 10.3109/17549501003746160. PMID 20433342
- [Background] Youmans SR, Youmans GL, Stierwalt JA. Differences in tongue strength across age and gender: is there a diminished strength reserve? Dysphagia. 2009 Mar;24(1):57-65. doi: 10.1007/s00455-008-9171-2. Epub 2008 Aug 9. PMID 18690406